CLINICAL TRIAL: NCT01011712
Title: The Natural History of Severe Viral Infections and Characterization of Immune Defects
Brief Title: The Natural History of Severe Viral Infections and Characterization of Immune Defects in Patients Without Known Immunocompromise
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100014; 10-I-0014
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-11-26

CONDITIONS: EBV; HSV; VZV; HPV; CMV
Keywords: Genetics; Virus; Defense; Immunity; Immunodeficiency; Natural History; Respiratory Viruses; Herpesvirus; Cytomegalovirus; Human Papillomavirus; Adenovirus
MeSH Terms: conditions — Virus Diseases; Immunologic Deficiency Syndromes; Herpes Simplex; Adenoviridae Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: patients without known or not fully characterized immunodeficiency, who have severe, persistent, or treatment-refractory viral infections

SUMMARY:
Background:

* Infections caused by viruses are common causes of illnesses: the common cold, many ear infections, sore throats, chicken pox, and the flu are caused by different viruses. Usually, these illnesses last only few days or, at most, a few weeks. Some virus infections like influenza are cleared from the body, and others such as the chicken pox virus remain in the body in an inactive state. However, some people may become quite ill when they are infected with a particular virus, possibly because part of their immune system does not respond properly to fight the virus.
* Researchers have discovered some reasons why a person may not be able to clear an infection caused by a virus. Some persons have changes in the genes that involve the immune system that result in the inability to properly control infection with a particular virus. Identifying changes in genes that involve the immune system should help scientists better understand how the immune system works to protect people from infection and may help develop new therapies.

Objectives:

* To study possible immune defects that may be linked to a particular severe viral infection.
* To determine if identified immune defects are genetic in origin.

Eligibility:

* Individuals of any age who have or have had a diagnosis of a virus infection that physicians consider to be unusually severe, prolonged, or difficult to treat.
* Relatives of the participants with a severe viral infection may also participate in the study. We will use their blood and/or skin specimens to try to determine if identified immune defects are hereditary.

Design:

* Prior to the study, the participant's doctor will give researchers the details of the infection, along with medical records for review. Eligible participants will be invited to the NIH Clinical Center for a full evaluation as an outpatient or inpatient.
* At the Clinical Center, participants will be treated with the best available therapy for the particular viral infection, and researchers will monitor how the infection responds to the treatment.
* Researchers will take intermittent blood samples and conduct other tests (such as skin biopsies) to evaluate the immune system. - During and after the illness, researchers will conduct follow-up visits to determine the course of infection and response to therapy.

DETAILED DESCRIPTION:
Viral infections in the normal host are usually self-limited as the innate and acquired immune systems mount successful antiviral responses. However, in some instances, apparently immunocompetent persons manifest infections with viruses that would otherwise be observed only in severely immunocompromised hosts. For example, cases of herpes simplex virus (HSV) encephalitis, esophagitis orgastritis, cytomegalovirus (CMV) colitis, adenovirus hepatitis or pneumonitis, recurrent or persistent skin infections caused by HSV or varicella zoster virus (VZV), severe warts caused by human papillomavirus (HPV), recurrent respiratory papillomatosis caused by HPV, severe influenza or respiratory syncytial virus pneumonia, and progressive multifocal leukoencephalopathy (PML) due to JC polyomavirus have been described in apparently immunocompetent patients. While a variety of case reports have described severe viral infections in immunocompetent hosts, the pathogenesis of the vast majority of these cases is not understood, and therapy can be unsuccessful.

In this protocol, we will evaluate patients without known immunocompromise, who have severe, persistent, or treatment-refractory viral infections caused by herpesviruses, adenoviruses, polyoma viruses, papillomaviruses, or other viral infections. We will investigate whether certain host or virologic factors predispose these individuals to severe disease. We will also determine the usefulness of various microbiologic tests (e.g., cultures, serology, molecular assays) for following the course of infection in these patients. The physicians in the Clinical Center will provide optimal therapy for these patients, as part of standard of care. Identification of virologic or host factors that predispose these patients to severe viral infections may have important implications for elucidating the pathogenesis of infection and for the development of novel therapies.

ELIGIBILITY:
* INCLUSION CRITERIA:

(Participants)

Participants must meet all the following inclusion criteria in order to participate in this study:

1. Children or adults (regardless of age) with a definitively diagnosed severe or unusual viral infection, including but not limited to infections caused by herpesviruses (HSV-1, HSV-2, CMV, EBV, VZV, HHV-6, HHV-7, HHV-8), human papillomavirus (e.g., severe recalcitrant warts), adenovirus, calicivirus (e.g. norovirus), polyomavirus (such as JC virus and BK virus), or influenza virus. Viral infections that would be considered opportunistic-like , such as herpesvirus esophagitis, herpesvirus encephalitis, CMV colitis, or progressive multifocal leukoencephalopathy (caused by the JC polyoma virus) will be of particular interest in this protocol.

   OR

   Children or adults with a well-documented prior, severe, persistent, or treatment-refractory viral infection(s), who have clinically recovered from the viral infection.
2. Ongoing care by a referring physician.
3. Willingness to allow storage of blood and tissue samples for future analyses.

(Relatives)

Relatives (2 years or above) may be recruited and enrolled to improve interpretation of genetic results, to expand the phenotype of the suspected or confirmed inborn error of immunity in the proband with severe viral infection, and to understand the co-factors in affected and/or unaffected family members that may influence variable expressivity and penetrance of viral infections in inborn errors of immunity.

1. Males and females will be accepted.
2. Relatives may either be healthy or have features concerning for an inborn error of immunity including, but not limited to, autoimmunity, severe atopy, other forms of immune-dysregulation, or severe or unusual infections. While the enrolled proband must have a current or prior severe or unusual viral infection, family members who are suspected to have an inborn error of immunity do not need to have a history of severe or unusual viral infection in the presence of other features suspicious for inborn errors of immunity.
3. Adult relatives or the guardians of minor relatives must be willing and capable of providing informed consent after review of protocol procedures that are described in the consent form with an appropriate study team member.
4. Participating relatives agree to have blood stored for future studies of the immune system.

EXCLUSION CRITERIA:

Participants meeting any of the following exclusion criteria at baseline will be excluded from study participation:

1. Patients with previously diagnosed conditions associated with acquired or iatrogenic immunodeficiency and/or immunosuppresion (e.g., a history of HIV infection, a positive test for HIV, chemotherapy or high dose glucocorticoids). Patients on immunosuppression and/or immunomodulatory therapy for the treatment of conditions that may be attributable to an underlying inborn error of immunity may be included in the study at the discretion of the PI or their designee.
2. Women who are pregnant.
3. Any condition or major comorbidity that the study investigators believe will compromise the patient's ability to comply with the requirements of the study.

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be drawn from referrals from the Clinical Center staff, physicians at outside medical facilities, and self-referrals. Patients or relatives who meet the inclusion and/or exclusion criteria, but who are not able to travel to the NIH Clinical Center, may be enrolled in the study and will be evaluated for immune defects using mailed-in blood samples or clinical specimens (i.e. previously obtained biopsy specimens).
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2009-10-01 (Actual)

PRIMARY OUTCOMES:
To find immune and/or genetic defects that predispose individuals to severe or unusual viral infections. | 10 years
  Patients under immune and genetic testing.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica R Durkee-Shock, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data generated by CLIA certified tests, such as whole exome sequencing results and numbers of immune cells, will be made available to the participant on this protocol.
Supporting Information: ICF
Time Frame: Whole exome sequencing results will be available approximately within 6 months to 1 year and if abnormal results are found they will be discussed by a genetics counselor with participants. Results from the Clinical Center Laboratory will be available within one to two weeks and will be discussed by the study team.
Access Criteria: IPD will be shared with the patient or in the case of children the parent who signed the consent as well as the child if they are felt to be mature enough to understand the results. IPD will also be discussed with the study team. If collaborations are initiated the samples will be coded so that the collaborator does not know the names of the patients.

REFERENCES:
- [Background] Dropulic LK, Ali MA, Ombrello AK, Cohen JI. Periodic Illness Associated With Epstein-Barr Virus: A New Diagnosis After a 22-Year Follow-up. Clin Infect Dis. 2016 Jun 15;62(12):1613-4. doi: 10.1093/cid/ciw197. Epub 2016 Mar 29. No abstract available. PMID 27025823
- [Background] Mace EM, Hsu AP, Monaco-Shawver L, Makedonas G, Rosen JB, Dropulic L, Cohen JI, Frenkel EP, Bagwell JC, Sullivan JL, Biron CA, Spalding C, Zerbe CS, Uzel G, Holland SM, Orange JS. Mutations in GATA2 cause human NK cell deficiency with specific loss of the CD56(bright) subset. Blood. 2013 Apr 4;121(14):2669-77. doi: 10.1182/blood-2012-09-453969. Epub 2013 Jan 30. PMID 23365458
- [Background] Dropulic LK, Cohen JI. Severe viral infections and primary immunodeficiencies. Clin Infect Dis. 2011 Nov;53(9):897-909. doi: 10.1093/cid/cir610. Epub 2011 Sep 29. PMID 21960712
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2010-I-0014.html